CLINICAL TRIAL: NCT02097186
Title: Preconditioning Shields Against Vascular Events in Surgery: A Multi-centre Feasibility Trial of Preconditioning Against Adverse Events in Major Vascular Surgery (Preconditioning-SAVES)
Brief Title: Preconditioning Shields Against Vascular Events in Surgery
Acronym: SAVES-F
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mid Western Regional Hospital, Ireland (Other)
Responsible Party: Principal Investigator, Professor Stewart Walsh, Prefessor Stewart Walsh, Mid Western Regional Hospital, Ireland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SAVES-F
Record Dates: First submitted 2014-03-24; First posted 2014-03-26 (Estimated); Last update posted 2014-12-12 (Estimated); Status verified 2014-12

CONDITIONS: Abdominal Aortic Aneurysm; Carotid Atherosclerosis; Critical Lower Limb Ischaemia
Keywords: Vascular disease; Open aortic aneurysm repair; Endovascular aneurysm repair; Carotid endartrectomy; Lower limb surgical revascularisation; Major lower limb amputation
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Carotid Artery Diseases; Vascular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Remote ischaemic preconditioning (Experimental): Remote ischaemic preconditioning will be performed in the same manner as several previous trials. Immediately after induction of anaesthesia, a standard, CE-approved blood pressure cuff will be placed around one arm of the patient. It will then be inflated to a pressure of 200mmHg for 5 minutes. For patients with a systolic blood pressure >185mmHg, the cuff will be inflated to at least 15mmHg above the patient's systolic blood pressure. The cuff will then be deflated and the arm allowed reperfuse for 5 minutes. This will be repeated so that each patient receives a total of 4 ischaemia-reperfusion cycles. In all other respects, the procedure and peri-operative care will follow the routine practices of the surgeons and anaesthetists involved.
  Interventions: Procedure: Remote ischaemic preconditioning
- Control to remote preconditioning group (No Intervention): Patients randomised to this group will receive routine pre-operative, peri-operative and post operative care.

INTERVENTIONS:
Procedure: Remote ischaemic preconditioning — Ischaemic preconditioning is a phenomenon whereby a brief period of non-lethal ischaemia in a tissue renders it resistant to the effects of a subsequent much longer ischaemic insult. Remote ischaemic preconditioning works on the theory that brief ischaemia in one tissue could confer protection on distant organs.
  Other Names: RIPC
  Arms: Remote ischaemic preconditioning

SUMMARY:
Major vascular surgery involves operations to repair swollen blood vessels, clear debris from blocked arteries or bypass blocked blood vessels. Patients with these problems are a high-risk surgical group as they have generalized blood vessel disease. These puts them at risk of major complications around the time of surgery such as heart attacks , strokes and death. The mortality following repair of a swollen main artery in the abdomen is about 1 in 20. This contrasts poorly with the 1 per 100 risk of death following a heart bypass. Simple and cost-effective methods are needed to reduce the risks of major vascular surgery. Remote ischaemic preconditioning (RIPC) may be such a technique. To induce RIPC, the blood supply to muscle in the patient's arm is interrupted for about 5 minutes. It is then restored for a further five minutes. This cycle is repeated three more times. The blood supply is interrupted simply by inflating a blood pressure cuff to maximum pressure. This repeated brief interruption of the muscular blood supply sends signals to critical organs such as the brain and heart, which are rendered temporarily resistant to damage from reduced blood supply. Several small randomized clinical trials in patients undergoing different types of major vascular surgery have demonstrated a potential benefit. This large, multi-centre trial aims to determine whether RIPC can reduce complications in routine practice.

DETAILED DESCRIPTION:
The demand for major vascular surgery is increasing [1]. Patients requiring procedures such as aortic aneurysm repair, carotid endarterectomy, lower limb surgical re-vascularisation and major lower limb amputation for end-stage vascular disease constitute a high-risk surgical cohort. Peri-operative complications such as myocardial infarction, cerebrovascular accident, renal failure and death are common [2,3]. Multiple potential mechanisms may result in these complications. For example, myocardial injury may result from systemic hypotension leading to reduced flow across a tight coronary artery stenosis or, alternatively, it may arise due to acute occlusion when an unstable plaque ruptures. Most strategies aimed at peri-operative risk reduction target a single potential mechanism. For example, beta-blockade may prevent myocardial injury due to overwork, but cannot prevent acute coronary occlusion. There is a requirement for a simple, effective intervention that protects tissues against injury via multiple different mechanisms. Remote ischemic preconditioning (RIPC) may be suitable.

Ischemic preconditioning is a phenomenon whereby a brief period of non-lethal ischemia in a tissue renders it resistant to the effects of a subsequent much longer ischaemic insult. It was first described in the canine heart [4]. Subsequent clinical trials showed that ischemic preconditioning reduced heart muscle damage following coronary artery bypass grafting [5] and liver dysfunction following hepatic resection [6]. Following cardiac surgery, it is associated with a reduction in critical care stay, arrhythmias and inotrope use [7]. However, ischemic preconditioning requires direct interference with the target tissues' blood supply, limiting its clinical utility. Further experimental work suggested that brief ischemia in one tissue, such as the kidneys, could confer protection on distant organs such as the heart [8]. A similar effect was observed after transient skeletal muscle ischemia [9-11]. This effect is referred to as 'preconditioning at a distance' or 'remote ischemic preconditioning' (RIPC).

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years
* Patient willing to give full informed consent for participation
* Patients undergoing elective carotid endarterectomy or
* Patients undergoing open abdominal aortic aneurysm repair or
* Patients undergoing endovascular abdominal aneurysm repair or
* Patients undergoing surgical lower limb revascularisation (suprainguinal or infrainguinal)

Exclusion Criteria:

* Pregnancy
* Significant upper limb peripheral arterial disease
* Previous history of upper limb deep vein thrombosis
* Patients on glibenclamide or nicorandil (these medications may interfere with RIPC) Patients with an estimated pre-operative glomerular filtration rate < 30mls/min/1.73m2
* Patients with a known history of myocarditis, pericarditis or amyloidosis
* Patients with an estimated pre-operative glomerular filtration rate < 30mls/min/1.73m2.
* Patients with severe hepatic disease defined as an international normalised ratio >2 in the absence of systemic anticoagulation
* Patients with severe respiratory disease (for the trial, defined as patients requiring home oxygen therapy)
* Patients previously enrolled in the trial representing for a further procedure
* Patients with previous axillary surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2014-04; Primary Completion 2016-04 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Serum troponin levels | 3 days
  The trial is intended to pragmatically evaluate the potential of RIPC to improve clinical outcomes among patients undergoing major vascular surgery in routine clinical practice. For the pilot trial, a surrogate marker of efficacy will be used, namely serum troponin I levels. The primary efficacy outcome will be a comparison of the proportion of patients in each arm of the trial who develop a serum troponin level in excess of the upper limit of normal in the first three post-operative days.

SECONDARY OUTCOMES:
Composite Major Adverse Clinical Events | 30 day
  The primary endpoint for the trial will be Major Adverse Clinical Events. This is a composite endpoint comprising any of: cardiovascular death, myocardial infarction, new onset arrhythmia requiring treatment, cardiac arrest, congestive cardiac failure, cerebrovascular accident, renal failure requiring renal replacement therapy, mesenteric ischaemia requiring intervention or biopsy proven ischaemic colitis, urgent cardiac revascularisation. All participants will undergo a serum troponin levels and 12-lead electrocardiogram on the second post-operative day to screen for silent peri-operative myocardial infarction. Trial ECGs and troponin levels will be interpreted by a blinded trial cardiologist.
Duration of post-operative hospital stay | 30 day
  The duration of hospital stay and ITU stay have a major impact on health service resource utilisation, and are factors which can be influenced by surgery.
Duration of intensive care unit stay | 30 day
  The duration of hospital stay and ITU stay have a major impact on health service resource utilisation, and are factors which can be influenced by surgery.
Unplanned critical care unit admission | 30 day
  The duration of hospital stay and ITU stay have a major impact on health service resource utilisation, and are factors which can be influenced by surgery.
Acute kidney injury score in first three peri-operative days | 3 days
  The Acute Kidney Injury Score will be calculated over the first three peri-operative days. Creatinine will be measured daily as part of routine care. Urine volumes will be calculated from the fluid balance charts maintained as part of usual care.
Post-operative complications | 30 day
  Postoperative complications will be recorded and results from both groups compared.
Mortality | 1 year
  Death within one year of surgery will be determined by contacting the patient's general practitioner.
Cardiac or cerebral event | 1 year
  Major adverse cardiac or cerebral event (myocardial infarction, cardiac death, cerebrovascular accident) within 1 year of surgery will be determined by contacting the patient's general practitioner for details.
Acute upper limb ischaemia | 24 hours post-operatively
  Acute upper limb ischaemia - This is defined as the development of ischaemia in the arm used for the preconditioning stimulus requiring systemic anti-coagulation, radiological intervention or surgical intervention. The arm will be assessed at the end of surgery to identify if ischaemia is present.
Acute upper limb deep vein thrombosis | 10 days
  Acute upper limb deep vein thrombosis - This is defined as the development of thrombus within the subclavian, axillary or brachial vein, which may develop up to 10 days post procedure, confirmed in duplex ultrasound and in the same arm as used for the RIPC stimulus.
Serial troponin I results | 3 days
  A comparison of the area under the curve of serial troponin I

OTHER OUTCOMES:
Acceptability of RIPC to patients | 6 weeks
  For patients, particularly those undergoing regional anaesthesia rather than general, the intervention may be burdensome and uncomfortable which may negatively impact upon likely adoption of this intervention into routine practice.In order to explore these potential issues, this feasibility trial will include a qualitative evaluation of acceptability to patients together with a qualitative evaluation of any perceived barriers to implementation. This evaluation will take the form of a semi-structured phone interview.
Acceptability and barriers to implementation among healthcare professionals. | 24 months
  Healthcare professionals at participating practices will be asked to complete a self-administered electronic questionnaire at the end of the study period. The questionnaire will elicit data on profession and practice details, their perceived experience of trial involvement, and open-ended questions to elicit information regarding attitudes to trial involvement, willingness to recruit participants, difficulties that arose during the trial and potential barriers to further research or routine clinical use of the trial intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Stewart R Walsh, Mch FRCS, Principal Investigator — Mid Western Regional Hospital and University of Limerick
Locations (6):
- Ireland (6):
  - Cork University Hospital, Cork, Cork
  - Beaumont Hospital, Dublin, Dublin
  - St James's Hospital, Dublin, Dublin
  - University Hospital Limerick (AKA MidWestern Regional Hospital), Limerick, Limerick
  - Waterford Regional Hospital, Waterford, Waterford
  - University Hospital Galway, Galway

REFERENCES:
- [Background] Anderson PL, Gelijns A, Moskowitz A, Arons R, Gupta L, Weinberg A, Faries PL, Nowygrod R, Kent KC. Understanding trends in inpatient surgical volume: vascular interventions, 1980-2000. J Vasc Surg. 2004 Jun;39(6):1200-8. doi: 10.1016/j.jvs.2004.02.039. PMID 15192558
- [Background] Chambers BR, Donnan GA. Carotid endarterectomy for asymptomatic carotid stenosis. Cochrane Database Syst Rev. 2005 Oct 19;2005(4):CD001923. doi: 10.1002/14651858.CD001923.pub2. PMID 16235289
- [Background] Greenhalgh RM, Brown LC, Kwong GP, Powell JT, Thompson SG; EVAR trial participants. Comparison of endovascular aneurysm repair with open repair in patients with abdominal aortic aneurysm (EVAR trial 1), 30-day operative mortality results: randomised controlled trial. Lancet. 2004 Sep 4-10;364(9437):843-8. doi: 10.1016/S0140-6736(04)16979-1. PMID 15351191
- [Background] Murry CE, Jennings RB, Reimer KA. Preconditioning with ischemia: a delay of lethal cell injury in ischemic myocardium. Circulation. 1986 Nov;74(5):1124-36. doi: 10.1161/01.cir.74.5.1124. PMID 3769170
- [Background] Jenkins DP, Pugsley WB, Alkhulaifi AM, Kemp M, Hooper J, Yellon DM. Ischaemic preconditioning reduces troponin T release in patients undergoing coronary artery bypass surgery. Heart. 1997 Apr;77(4):314-8. doi: 10.1136/hrt.77.4.314. PMID 9155608
- [Background] Clavien PA, Selzner M, Rudiger HA, Graf R, Kadry Z, Rousson V, Jochum W. A prospective randomized study in 100 consecutive patients undergoing major liver resection with versus without ischemic preconditioning. Ann Surg. 2003 Dec;238(6):843-50; discussion 851-2. doi: 10.1097/01.sla.0000098620.27623.7d. PMID 14631221
- [Background] Walsh SR, Tang TY, Kullar P, Jenkins DP, Dutka DP, Gaunt ME. Ischaemic preconditioning during cardiac surgery: systematic review and meta-analysis of perioperative outcomes in randomised clinical trials. Eur J Cardiothorac Surg. 2008 Nov;34(5):985-94. doi: 10.1016/j.ejcts.2008.07.062. Epub 2008 Sep 9. PMID 18783958
- [Background] Przyklenk K, Bauer B, Ovize M, Kloner RA, Whittaker P. Regional ischemic 'preconditioning' protects remote virgin myocardium from subsequent sustained coronary occlusion. Circulation. 1993 Mar;87(3):893-9. doi: 10.1161/01.cir.87.3.893. PMID 7680290
- [Background] Birnbaum Y, Hale SL, Kloner RA. Ischemic preconditioning at a distance: reduction of myocardial infarct size by partial reduction of blood supply combined with rapid stimulation of the gastrocnemius muscle in the rabbit. Circulation. 1997 Sep 2;96(5):1641-6. doi: 10.1161/01.cir.96.5.1641. PMID 9315559
- [Background] Kharbanda RK, Mortensen UM, White PA, Kristiansen SB, Schmidt MR, Hoschtitzky JA, Vogel M, Sorensen K, Redington AN, MacAllister R. Transient limb ischemia induces remote ischemic preconditioning in vivo. Circulation. 2002 Dec 3;106(23):2881-3. doi: 10.1161/01.cir.0000043806.51912.9b. PMID 12460865
- [Background] Oxman T, Arad M, Klein R, Avazov N, Rabinowitz B. Limb ischemia preconditions the heart against reperfusion tachyarrhythmia. Am J Physiol. 1997 Oct;273(4):H1707-12. doi: 10.1152/ajpheart.1997.273.4.H1707. PMID 9362234
- [Derived] Healy D, Clarke-Moloney M, Gaughan B, O'Daly S, Hausenloy D, Sharif F, Newell J, O'Donnell M, Grace P, Forbes JF, Cullen W, Kavanagh E, Burke P, Cross S, Dowdall J, McMonagle M, Fulton G, Manning BJ, Kheirelseid EA, Leahy A, Moneley D, Naughton P, Boyle E, McHugh S, Madhaven P, O'Neill S, Martin Z, Courtney D, Tubassam M, Sultan S, McCartan D, Medani M, Walsh S. Preconditioning Shields Against Vascular Events in Surgery (SAVES), a multicentre feasibility trial of preconditioning against adverse events in major vascular surgery: study protocol for a randomised control trial. Trials. 2015 Apr 23;16:185. doi: 10.1186/s13063-015-0678-1. PMID 25903752